CLINICAL TRIAL: NCT03593720
Title: Glans Size in Hypospadias Compared to Normal
Status: Completed | Type: Observational
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Barry Kogan, MD, Professor of Surgery and Pediatrics, Albany Medical College
Other Study IDs: AMC5152
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Hypospadias; Surgery Non Hypospadias
Keywords: hypaspadias
MeSH Terms: conditions — Hypospadias | interventions — Weights and Measures; Working Conditions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypospadias: Patients with hypospadias
  Interventions: Procedure: Measurement in Office; Procedure: Measurement in OR
- Control: Patients without hypospadias
  Interventions: Procedure: Measurement in OR

INTERVENTIONS:
Procedure: Measurement in Office — Penile length and glans size in 3 dimensions
  Groups: Hypospadias
Procedure: Measurement in OR — Penile length and glans size in 3 dimensions

SUMMARY:
The investigator will collect data on penile and glans size by age, weight and ethnicity in both patients undergoing routine urological surgery and hypospadias surgery.

DETAILED DESCRIPTION:
After obtaining informed consent , the investigator will measure stretched penile length and glans size in 3 dimensions (length, width, height) in the office on patients with hypospadias, as well as at the time of operation, after the induction of anesthesia. Patients undergoing hypospadias surgery will be considered study subjects. If the patient was given pre-operative testosterone as part of the current standard of care, this will be noted and the measurements taken at each pre-operative office visit will be recorded. The investigator will also record corrected age, weight in kilograms and ethnicity as identified by the family.

Control patients will be those male patients undergoing non-hypospadias urological surgery (hernia repair, orchiopexy, circumcision, re-circumcision) with a normal penis, the investigator will perform a single intra-operative measurement of the same glans and penile variables after induction of anesthesia and prior to the start of their genital surgery. Again, age, weight and ethnicity will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery for hypospadias
* Patients undergoing any urologic surgery other than hypospadias

Exclusion Criteria:

* other penile abnormalities (Hidden penis, penoscrotal wedding/transposition, chordee without hypospadias, penile torsion, etc.)
* Undergoing other penile procedures (penoplasty, chordee repair, penile detorsion, etc.)

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The source of subjects will be patients examined in the Pediatric Urology clinic and operating room. In contemporary practice, most hypospadias surgery is conducted at less than two years of age. Total of patients enrolled will be 90, with 45 in each the control and study group. The study population are patients undergoing surgery for hypospadias and the control population are patients undergoing any urologic surgery other than hypospadias.
Sampling Method: Non-Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2024-12-29 (Actual); Study Completion 2024-12-29 (Actual)

PRIMARY OUTCOMES:
Difference in glans size between hypospadias patients and those without hypospadias | 6 months
  The investigator will prospectively collect data on glans size by age, weight and ethnicity in both patients undergoing routine urological surgery and hypospadias surgery

SECONDARY OUTCOMES:
Difference in penile length between hypospadias patients and those without hypospadias | 6 months
  The investigator will prospectively collect data on penis length by age, weight and ethnicity in both patients undergoing routine urological surgery and hypospadias surgery
Track penile and glans growth curves in both cohorts | 24 months
  The investigator will prospectively track penile and glans growth over time to develop longitudinal growth curves in both cohorts
Determine the effect of testosterone on penile and glans growth in hypospadias | 24 months
  The investigator will measure the glans size and penile length of patients who receive testosterone for small glans size before and after administration in order to determine the effect of testosterone administration.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Kogan, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical College, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Babu R. Glans meatus proportion in hypospadias versus normal: does marking reference points impact outcome? J Pediatr Urol. 2014 Jun;10(3):459-62. doi: 10.1016/j.jpurol.2013.11.008. Epub 2013 Nov 28. PMID 24332704
- [Background] Bush NC, DaJusta D, Snodgrass WT. Glans penis width in patients with hypospadias compared to healthy controls. J Pediatr Urol. 2013 Dec;9(6 Pt B):1188-91. doi: 10.1016/j.jpurol.2013.05.004. Epub 2013 Jun 12. PMID 23768835
- [Background] Bush NC, Villanueva C, Snodgrass W. Glans size is an independent risk factor for urethroplasty complications after hypospadias repair. J Pediatr Urol. 2015 Dec;11(6):355.e1-5. doi: 10.1016/j.jpurol.2015.05.029. Epub 2015 Aug 13. PMID 26320396
- [Background] Malik RD, Liu DB. Survey of pediatric urologists on the preoperative use of testosterone in the surgical correction of hypospadias. J Pediatr Urol. 2014 Oct;10(5):840-3. doi: 10.1016/j.jpurol.2014.02.008. Epub 2014 Mar 18. PMID 24726783
- [Background] Babu R, Chakravarthi S. The role of preoperative intra muscular testosterone in improving functional and cosmetic outcomes following hypospadias repair: A prospective randomized study. J Pediatr Urol. 2018 Feb;14(1):29.e1-29.e6. doi: 10.1016/j.jpurol.2017.07.009. Epub 2017 Aug 12. PMID 28844754
- [Background] Chua ME, Gnech M, Ming JM, Silangcruz JM, Sanger S, Lopes RI, Lorenzo AJ, Braga LH. Preoperative hormonal stimulation effect on hypospadias repair complications: Meta-analysis of observational versus randomized controlled studies. J Pediatr Urol. 2017 Oct;13(5):470-480. doi: 10.1016/j.jpurol.2017.06.019. Epub 2017 Jul 29. PMID 28939350
- [Background] Rynja SP, de Jong TPVM, Bosch JLHR, de Kort LMO. Testosterone prior to hypospadias repair: Postoperative complication rates and long-term cosmetic results, penile length and body height. J Pediatr Urol. 2018 Feb;14(1):31.e1-31.e8. doi: 10.1016/j.jpurol.2017.09.020. Epub 2017 Oct 27. PMID 29174377
- [Background] Van Praet C, Spinoit AF. Testosterone prior to hypospadias repair: No clear-cut benefit or reassurance regarding long-term safety. J Pediatr Urol. 2018 Feb;14(1):85-86. doi: 10.1016/j.jpurol.2017.11.006. Epub 2017 Nov 27. No abstract available. PMID 29248308
- [Background] Asgari SA, Safarinejad MR, Poorreza F, Asl AS, Ghanaie MM, Shahab E. The effect of parenteral testosterone administration prior to hypospadias surgery: A prospective, randomized and controlled study. J Pediatr Urol. 2015 Jun;11(3):143.e1-6. doi: 10.1016/j.jpurol.2014.12.014. Epub 2015 Mar 12. PMID 25837705
- [Background] Paiva KC, Bastos AN, Miana LP, Barros Ede S, Ramos PS, Miranda LM, Faria NM, Avarese de Figueiredo A, de Bessa J Jr, Netto JM. Biometry of the hypospadic penis after hormone therapy (testosterone and estrogen): A randomized, double-blind controlled trial. J Pediatr Urol. 2016 Aug;12(4):200.e1-6. doi: 10.1016/j.jpurol.2016.04.013. Epub 2016 May 26. PMID 27321554
- [Background] Puri A, Sikdar S, Prakash R. Pediatric Penile and Glans Anthropometry Nomograms: An Aid in Hypospadias Management. J Indian Assoc Pediatr Surg. 2017 Jan-Mar;22(1):9-12. doi: 10.4103/0971-9261.194610. PMID 28082769